Minimally Invasive Treatment Approach for Early Childhood Caries Using Silver Diammine Fluoride and NaF With Functionalized Tricalcium Phosphate and Their Effects on Oral Health Related Quality of Life: A Pragmatic RCT

## Subject Information and Consent Form (Signature Page) Research Title: Researcher's Name:

To become a part this study, you or your legal representative must sign this page. By signing this page, I am confirming the following:

- I have read all of the information in this Patient Information and Consent Form including any information regarding the risk in this study and I have had time to think about it.
- All of my questions have been answered to my satisfaction.
- I voluntarily agree to be part of this research study, to follow the study procedures, and to provide necessary information to the doctor, nurses, or other staff members, as requested.
- I may freely choose to stop being a part of this study at anytime.
- I have received a copy of this Participant Information and Consent Form to keep for myself.

| Participant Name | _ |
|-------------------------------------------------------|-----------------|
| Participant I.C No | _ |
| Signature of Participant or Legal Representative | Date (dd/MM/yy) |
| Name of Individual Conducting Consent Discussion | _ |
| Signature of Individual Conducting Consent Discussion | Date (dd/MM/yy) |
| Name & Signature of Witness | Date (dd/MM/yy) |

Note: i) All participants who are involved in this study will not be covered by insurance.

## Subject Information and Consent Form (Signature Page – Genetic Sample) Research Title: Researcher's Name:

To become a part this study, you or your legal representative must sign this page. By signing this page, I am confirming the following:

- I have read all of the information in this Patient Information and Consent Form including any information regarding the risk in this study and I have had time to think about it.
- All of my questions have been answered to my satisfaction.
- I voluntarily agree to be part of this research study, to follow the study procedures, and to provide necessary information to the doctor, nurses, or other staff members, as requested.
- I may freely choose to stop being a part of this study at anytime.
- I have received a copy of this Participant Information and Consent Form to keep for myself.

| Participant Name | |
|-------------------------------------------------------|-----------------|
| Participant I.C No. | |
| Signature of Participant or Legal Representative | Date (dd/MM/yy) |
| Name of Individual conducting Consent Discussion | |
| Signature of Individual Conducting Consent Discussion | Date (dd/MM/yy) |
| Name & Signature of Witness | Date (dd/MM/yy) |

Note: i) All participants who are involved in this study will not be covered by insurance.

ii) Excess samples from this research will not be used for other reasons and will be destroyed with the consent from the Human Research Ethics Committee, USM.

| Participant's Material Publication Consent Form Signature Page | |
|---|---|
| Research 1 | Title: |
| Researche | r's Name: |
| To become | a part this study, you or your legal representative must sign this page. |
| By signing t | his page, I am confirming the following: |
| • | I understood that my name will not appear on the materials published and there have been efforts to make sure that the privacy of my name is kept confidential although the confidentiality is not completely guaranteed due to unexpected circumstances. |
| • | I have read the materials or general description of what the material contains and reviewed all photographs and figures in which I am included that could be published. |
| | I have been offered the opportunity to read the manuscript and to see all materials in which I am included, but have waived my right to do so. |
| • | All the published materials will be shared among the medical practitioners, scientists and journalist world wide. |
| • | The materials will also be used in local publications, book publications and accessed by many local and international doctors world wide. |
| • | I hereby agree and allow the materials to be used in other publications required by other publishers with these conditions: |
| • | The materials will not be used as advertisement purposes nor as packaging materials. |
| • | The materials will not be used out of contex — i.e.: Sample pictures will not be used in an article which is unrelated subject to the picture. |
| Participant | |
| Participant | I.C No. Participant's Signature Date (dd/MM/yy) |

Note: i) All participants who are involved in this study will not be covered by insurance.

Name and Signature of Individual

Conducting Consent Discussion

Date (dd/MM/yy)